CLINICAL TRIAL: NCT02392130
Title: A Prospective, Randomised, Investigator-Blinded, Vehicle-Controlled, Phase I Clinical Trial With Intra-Individual Comparison of Treatments to Assess the Potential of LEO 130852A Gel to Reduce Steroid Induced Skin Atrophy on Healthy Skin
Brief Title: A Clinical Trial to Assess the Potential of LEO 130852A Gel to Reduce Steroid Induced Skin Atrophy on Healthy Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SKAT-1129
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Skin Tissue Diseases; Connective Tissue Diseases
MeSH Terms: conditions — Connective Tissue Diseases | interventions — Clobetasol; Ointments

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Drug (Active Comparator): Clobetasol propionate 0.05% ointment
  Interventions: Drug: Clobetasol propionate 0.05% ointment
- Experimental Drug (Experimental): LEO 130852A gel 1%
  Interventions: Drug: LEO 130852A gel 1%
- Placebo Drug (Placebo Comparator): LEO 130852A placebo gel
  Interventions: Drug: LEO 130852A placebo gel

INTERVENTIONS:
Drug: Clobetasol propionate 0.05% ointment
  Arms: Active Drug
Drug: LEO 130852A gel 1%
  Arms: Experimental Drug
Drug: LEO 130852A placebo gel
  Arms: Placebo Drug

SUMMARY:
The purpose of this study is to assess the effect of LEO 130852A gel 1% in maintaining skin thickness in healthy skin treated with steroid.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 25 to 50 years old inclusive
* Healthy skin on volar arms with a hairless area sufficient for measurements

Exclusion Criteria:

* Clinical skin atrophy, telangiectasia or striae on volar arms
* Presence of any skin condition or colouration that would interfere with test sites or the response or assessment
* Fitzpatrick skin type IV - VI
* History or current evidence of infection, eczema or other relevant skin disease

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Skin thickness measured by sonography and histology | 4 weeks

SECONDARY OUTCOMES:
Clinical assessments measured by atrophy score | 4 weeks
Clinical assessments measured by telangiectasia score | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- bioskin GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en